CLINICAL TRIAL: NCT00003894
Title: Thalidomide vs. Placebo for Steroid Dependent or Refractory Chronic Graft vs. Host Disease (cGVHD) IND #42782
Brief Title: Thalidomide in Treating Patients With Chronic Graft-Versus-Host Disease Following Bone Marrow Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Barbara Bambech, MD, Roswell Park Cancer Institute
Model: Parallel | Purpose: Supportive Care
Other Study IDs: CDR0000067064; RPCI-RP-9809
Record Dates: First submitted 1999-11-01; First posted 2004-06-17 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Graft Versus Host Disease; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may interfere with the body's ability to recognize transplanted bone marrow cells as foreign and may help treat patients with graft-versus-host disease.

PURPOSE: Randomized phase II trial to study the effectiveness of thalidomide in treating patients who have chronic graft-versus-host disease following bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of thalidomide in patients with steroid dependent or refractory chronic graft vs host disease following an allogeneic bone marrow transplant. II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to the type of bone marrow transplant received (allogeneic vs matched unrelated donor) and type of chronic graft vs host disease (steroid dependent vs steroid refractory). Patients receive either oral thalidomide or placebo 2-4 times a day for 6 months. The drug is then tapered until stopped. If disease recurs, the drug may be restarted for a second 6 month course. The maximum duration of treatment is 18 months. Patients continue on steroid therapy, which is tapered during study therapy. If no response is seen after 8 weeks, patients may cross over to the other alternate drug. Patients are followed weekly for 1 month, then every month for 1 year.

PROJECTED ACCRUAL: A total of 36 patients (18 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed chronic graft vs host disease following an allogeneic bone marrow transplant (BMT) Greater than 100 days since BMT Must be receiving at least 1 mg/kg of prednisone or equivalent immunosuppression

PATIENT CHARACTERISTICS: Age: 3 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Radiotherapy: Not specified Surgery: Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1999-03; Primary Completion 2000-01 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (10):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Roswell Park Cancer Institute, Buffalo, New York
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center of the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin